CLINICAL TRIAL: NCT01253031
Title: Effects of Aging and Hearing Loss During Rapid Sound Processing
Brief Title: Working Memory Changes With Aging and Hearing Loss
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C6928-P
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Aging; Hearing Loss
Keywords: hearing loss; aging; short term memory; attentional blink
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1: young normal hearing
- Group 2: older normal hearing
- Group 3: older hearing impaired

SUMMARY:
Hearing loss is one of the most common health concerns affecting 1 in 3 Americans over 60 years of age rising to 1 in 2 for those over 85 years old. Contributions to hearing abilities provided by cognitive and memory processes are universally recognized as essential to adequate speech communication, but these processes are not well understood. Cognitive limitations in the ability to rapidly process sequential sounds occur with all listeners but may have more impact on older Veterans with and without hearing impairment. The purpose of this study is to examine and more thoroughly characterize the change in auditory working memory with hearing loss and increasing age. Young and older listeners with and without hearing loss will listen and report on two target sounds embedded in a stream of rapidly occurring sound. The investigators expect that older listeners without hearing loss will have more difficulty than young listeners but that older listeners with hearing impairment will have the most difficulty with this task even when the sounds they are listening to are adjusted to compensate for their hearing loss.

DETAILED DESCRIPTION:
The purpose of this pilot study is to understand how memory changes with aging and if failures of working memory during rapid sound processing may account for some of the speech perception difficulties reported by older Veteran listeners especially those with hearing loss. A period of processing interference (and limitation) has been identified during rapid auditory or visual processing. Specifically, when subjects are asked to report on two targeted events embedded in a rapid stream of distractor events, the ability to report on the second target is diminished when it occurs at an interval of approximately 200-400ms following the first target. This has been identified as a failure of working memory consolidation and is robust during both visual and auditory processing. Much is known about how the failure of working memory affects young normal hearing listeners but little is known of its effect on older listeners or listeners with hearing loss. A lengthened period of processing interference is very likely to be present among older listeners. This is important because speech is rapid and older listeners often report difficulty in auditory environments in which multiple speakers are present. Further, older listeners, who are more likely to have hearing loss, continue to report more problems hearing in noisy environments even with their hearing aids optimally functional. The presence of a prolonged period of processing interference in the auditory system could account for some of these complaints and, if more completely understood, could be remediated.

Up to 75 subjects, ages 18-30 and 60-75 years will be invited to participate. Subjects will undergo a complete audiological evaluation done to assign them into one of three arms/groups of up to15 subjects each. Arms will be composed of young subjects with normal hearing (YNH), older subjects with normal hearing (ONH) and older subjects with mild hearing impairment (OHI). Each subject will be asked to listen to between 18 and 26 non-overlapping tones each 30ms in duration followed by a 70ms silent interval. Target tones and tone complexes (T1 and T2) will be embedded in this stream. Sequences could contain (in equal probability) a) no target, b) T1 only, c) T2 only or d) both targets. At the end of each stream, the subject will be required to make an untimed judgment about whether the stream contained T1 (yes/no) and T2 (yes/no). This project is self-paced. The hypothesized findings are that young listeners without hearing impairment will have more difficulty reporting on T2 when it follows T1 by approximately 200-400ms than at any other interval. However, older listeners without hearing impairment will demonstrate a more prolonged period of interference (>400ms) with slightly poorer performance overall while older listeners with hearing impairment will have an even longer lasting period of processing interference and overall larger deficit (poorer performance) suggesting that increasing age and hearing impairment combine to reveal significant processing deficits for this group. These results would provide a much needed explanation of the ways in which rapid processing (precisely what speech is) is degraded by hearing impairment, aging, and a combination of the two.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age or 60-75 years of age
* Normal hearing or
* Mild to moderate hearing loss
* No major medical or memory problems

Exclusion Criteria:

* <24/30 on MMSE
* Conductive or mixed hearing loss.
* Hearing loss worse than 55dB in either ear.
* Taking medication known to alter concentration or alertness
* Inability to learn task after practice
* Major medical or psychological disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All populations meeting the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Time between targets (lag time) | At time of consent up to 2 weeks from consent
  The subjects will be trained to hear each target sound in a sequence of sounds. The target sounds will vary in terms of how closely they occur to each other. Closer (in time, also called lag time) targets will be harder to hear than far apart (in time) targets.

SECONDARY OUTCOMES:
Percent correct | At time of consent up to 2 weeks from consent

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn L Dille, PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States